CLINICAL TRIAL: NCT02009787
Title: Effect of Vitamin D and Statins on Plasma Lipid Profiles in Chinese Patients With Hypercholesterolemia
Brief Title: Efficacy Study of Vitamin D and Statins to Treat Hypercholesterolemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shi Yang (Other)
Responsible Party: Sponsor-Investigator, Shi Yang, Director of Geriatric Cardiology, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S2013-098-01
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Primary Hypercholesterolemia
Keywords: hypercholesterolemia; vitamin D; adjuvant therapy
MeSH Terms: conditions — Hypercholesterolemia | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D supplementation group (Experimental): drug: vitamin D3 tablets (Vigantoletten; Merck Pharma, Germany); the frequency: 2000 IU vitamin D3 tablets were taken daily; duration: 6 months.
  Interventions: Drug: vitamin D3 tablets
- Control group (Placebo Comparator): drug: placebo tablets; the frequency: 2000 IU placebo tablets were taken daily; duration: 6 months.
  Interventions: Drug: placebo tablets

INTERVENTIONS:
Drug: vitamin D3 tablets — 2000 IU vitamin D3 tablets were taken daily for 6 months
  Other Names: Vigantoletten; Merck Pharma, Germany
  Arms: Vitamin D supplementation group
Drug: placebo tablets — 2000 IU placebo tablets were taken daily for 6 months
  Arms: Control group

SUMMARY:
The investigators planned to research the effect of vitamin D supplementation as an adjuvant therapy for patients with hypercholesterolemia.

DETAILED DESCRIPTION:
Vitamin D is primarily generated in the skin, in response to direct absorption of ultraviolet B radiation. Vitamin D can also be obtained through fortified foods and oral supplements. Lipid abnormalities are common in the general population, and are regarded as a modifiable risk factor for cardiovascular disease. Recently low vitamin D status has been shown to be associated with increased risk of developing hyperlipidemia. Statins are normally the first-line therapy for hypercholesterolemia. It is also reported that vitamin D can improve serum lipid levels. However, its effects on hypercholesterolemia patients remain unclear. The investigators planned to determine the efficacy of combination therapy with statins and vitamin D in a cohort of hypercholesterolemia patients. This study may shed light as to whether oral vitamin D supplementation can be an adjunct therapy in hypercholesterolemia patients.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria were for hypercholesterolemia patients with the treatment of statins.

Exclusion Criteria:

The exclusion criteria were as follows: patients with chronic renal failure, chronic liver disease, bone disorders, and/or thyroid disorders. Patients were also excluded if they were taking vitamin D3 tablets or other lipid-regulating drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
a change in serum total cholesterol level | after 6 months of vitamin D supplementation
  The primary end point was a change in serum total cholesterol level after 6 months of vitamin D supplementation.

SECONDARY OUTCOMES:
a change in serum triglycerides level | after 6 months of vitamin D supplementation
  The change in serum triglycerides level was measured after 6 months of vitamin D supplementation.
differences in the incidences of treatment-emergent adverse events | after 6 months of vitamin D supplementation
  Treatment-emergent adverse events (TEAEs): hypercalcemia, renal insufficiency, constipation

CONTACTS AND LOCATIONS:
Overall Officials: Yu Tang Wang, M.D., Study Director — PLA General Hospital
Locations (1):
- PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Kendrick J, Targher G, Smits G, Chonchol M. 25-Hydroxyvitamin D deficiency is independently associated with cardiovascular disease in the Third National Health and Nutrition Examination Survey. Atherosclerosis. 2009 Jul;205(1):255-60. doi: 10.1016/j.atherosclerosis.2008.10.033. Epub 2008 Nov 11. PMID 19091317
- [Background] Botella-Carretero JI, Alvarez-Blasco F, Villafruela JJ, Balsa JA, Vazquez C, Escobar-Morreale HF. Vitamin D deficiency is associated with the metabolic syndrome in morbid obesity. Clin Nutr. 2007 Oct;26(5):573-80. doi: 10.1016/j.clnu.2007.05.009. Epub 2007 Jul 10. PMID 17624643
- [Background] Skaaby T, Husemoen LL, Pisinger C, Jorgensen T, Thuesen BH, Fenger M, Linneberg A. Vitamin D status and changes in cardiovascular risk factors: a prospective study of a general population. Cardiology. 2012;123(1):62-70. doi: 10.1159/000341277. Epub 2012 Sep 12. PMID 22986625
- [Background] Ponda MP, Dowd K, Finkielstein D, Holt PR, Breslow JL. The short-term effects of vitamin D repletion on cholesterol: a randomized, placebo-controlled trial. Arterioscler Thromb Vasc Biol. 2012 Oct;32(10):2510-5. doi: 10.1161/ATVBAHA.112.254110. Epub 2012 Sep 4. PMID 22947589
- [Result] Schwartz JB. Effects of vitamin D supplementation in atorvastatin-treated patients: a new drug interaction with an unexpected consequence. Clin Pharmacol Ther. 2009 Feb;85(2):198-203. doi: 10.1038/clpt.2008.165. Epub 2008 Aug 27. PMID 18754003
- [Derived] Qin XF, Zhao LS, Chen WR, Yin DW, Wang H. Effects of vitamin D on plasma lipid profiles in statin-treated patients with hypercholesterolemia: A randomized placebo-controlled trial. Clin Nutr. 2015 Apr;34(2):201-6. doi: 10.1016/j.clnu.2014.04.017. Epub 2014 May 2. PMID 24844869